CLINICAL TRIAL: NCT06016114
Title: Analysis of the Reservoir in Individuals Controlling HIV Infection
Acronym: ARCH
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ID 12241 - ARCH
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hiv
Keywords: HIV; Latency
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HIV-1 positive individuals (non-pregnant)
  Interventions: Diagnostic Test: HIV Latency Diagnostic Sampling
- Pregnant HIV-1 positive/negative individuals
  Interventions: Diagnostic Test: HIV Latency Diagnostic Sampling

INTERVENTIONS:
Diagnostic Test: HIV Latency Diagnostic Sampling — This intervention involves the collection of blood, lymph node, colon biopsy, and placental samples from individuals living with HIV (HIV controllers) and healthy controls. The goal is to investigate HIV latency by analyzing these biological samples to gain insights into the mechanisms and characteristics of latent HIV reservoirs. The sampling procedures will be conducted using minimally invasive techniques where appropriate, and the collected samples will undergo laboratory analysis for further study.

SUMMARY:
The aim of this study is the gain new insights into HIV latency in HIV controllers through extensive blood an tissue sampling (lymph node, colon biopsies, placenta) from 25 individuals living with HIV and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Elite Controllers: pVL<50 copies per ml for at least 12 months, treatment naive at the time of inclusion
* Viral controllers: pVL <2000 copies/ml; CD4>500/µL for at least two years, treatment naïve at the time of inclusion
* Long-term non-progressors: CD4>500/µL, pVL <10000 copies/ml, for at least 7 years, treatment naïve at the time of inclusion
* Post treatment controllers: on cART for at least 12 months; pVL <500 copies/ml for at least 2 years after treatment cessation .
* PLWH who received bone marrow transplant: people living with HIV who received a bone-marrow transplant for non-HIV related reasons

Exclusion Criteria:

* Current history of opportunistic infection (AIDS defining events as defined in category C of the CDC clinical classification), consisting of chronic HIV-1 infection.
* Evidence of active HBV infection (Hepatitis B surface antigen positive or HBV viral load positive in the past and no evidence of subsequent seroconversion (= HBV antigen or viral load negative and positive HBV surface antibody)).
* Evidence of active HCV infection (HCV antibody positive result within 60 days prior to study entry with positive HCV viral load or, if the HCV antibody result is negative, a positive HCV RNA result within 60 days prior to study entry).
* Current or known history of cardiomyopathy or significant ischemic or cerebrovascular disease.
* Current history of cancer.
* History of HIV-related thrombocytopenia.
* Any condition, including preexisting psychiatric and psychological disorders, which will in the opinion of the investigator interfere with the trial conduct or safety of the participant.
* Abnormal results of standard of care laboratory tests:

  1. Confirmed haemoglobin <11g/dl for women and <12 g/dl for men
  2. Confirmed platelet count <100 000/µl *
  3. Confirmed neutrophil count <1000/μl
  4. Confirmed AST and/or ALT >10xULN
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 60 days prior to entry.
* The following treatment will be prohibited three months before screening and during the study:

  1. immunosuppressive drugs (inclusive corticosteroids) except for drugs used for topical use.
  2. Immunomodulatory drugs including but not limited to Granulocyte-colony stimulating factors, Granulocyte-monocyte colony-stimulating factor, interleukin 2, 7 & 15.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-positive individuals (pregnant and non-pregnant) and pregnant HIV-negative individuals
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of total and intact HIV DNA and HIV RNA | 5 years
  Rainbow assay: multiplex digital PCR approach that combines five different HIV-1 regions to quantify total HIV-1 DNA and intact HIV-1 DNA simultaneously (Qiacuity dPCR platform, Qiagen).
  mutliplex digital PCR approach to quantify HIV RNA
Integration site analysis | 5 years
  HIV/host DNA junctions will be amplified using the Integration Site Loop Amplification (ISLA) assay, and resulting chimeric amplicons will be sequenced by Sanger.
Full-length HIV genome analysis | 5 years
  Full-Length Individual Proviral Sequencing (FLIPS) assay: nested PCR with Illumina MiSeq.
Epigenetic analysis | 5 years
  Methylation (bisulfite conversion) and chromatin accessibility (Assay for Transposase-Accessible Chromatin using sequencing)
Matched integration site and proviral sequencing | 5 years
  MIP-seq: captures full-length viral genome sequences in conjunction with its associated viral integration site
Proviral UMI-mediated Long-read Sequencing | 5 years
  HIV-PULSE: characterize the composition of the viral reservoir using long-read sequencing. Involves pre-amplifying individual proviral genomes using PCR and tagging them with dual UMIs, followed by long-range PCR amplification and long-read sequencing on the Oxford Nanopore MinION platform
Transcriptome analysis | 5 years
  * Bulk RNA sequencing on extracted RNA (Illumina Hiseq 2500 with 10-100 ng input of ribodepleted RNA)
  * Single cell RNA sequencing (10x genomics technology )
High dimensional phenotyping | 5 years
  CyTOF (mass cytometry, Fluidigm) combined with bioinformatics approach to extensively characterize the phenotype of latently infected cells
Immunohistochemistry, RNA- and DNA In Situ Hybridization | 5 years
  Immunochemistry will be used to study the expression of activation and exhaustion markers on tissues samples , while viral expression will be assessed through DNAScope and RNAScope technologies
Immunometabolic profile analysis | 5 years
  Mass spectrometry metabolomics will be used to study the immunometabolic profile of latently infected cells
Detection of translation-competent reservoirs | 5 years
  HIV-Flow assay: flow cytometry based assay using a combination of 2 antibodies targeting the p24 protein and allowing the detection of cells containing translation-competent viruses. p24+ cells detected by this assay can be sorted for downstream applications and further characterization of translation-competent reservoirs.
  The Simultaneous TCR Integration site and Provirus sequencing (STIP-seq) assay will be performed to sequence the proviral genome and matched integration sites of the translation-competent viruses, as well as phenotypic characterization and TCR sequencing of the host cell. characterization of translation-competent reservoirs.
Immunological analysis-FACS | 5 years
  Immunophenotyping by flow cytometric assays will be performed of different cells to assess the phenotype of innate immune cells, using FACS analysis.
Immunological analysis-ELISA | 5 years
  Immunophenotyping by flow cytometric assays will be performed of different cells to assess the phenotype of innate immune cells, using ELISA.
Microbiome monitoring | 5 years
  Gut microbiome will be analyzed in stool and colon biopsies using next-generation sequencing (NGS) of rRNA gene amplicons to identify bacteria at genus/species level

CONTACTS AND LOCATIONS:
Overall Officials: Linos Vandekerckhove, MD PhD, Principal Investigator — University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No